CLINICAL TRIAL: NCT01965951
Title: RESPONSE: Remediation of Spatial Neglect Trial
Brief Title: Remediation of Spatial Neglect Trial
Acronym: RESPONSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: Washington University School of Medicine (Other); VA Boston Healthcare System (U.S. Federal Agency); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-1004-13
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Acquired Brain Injury; Hemispatial Neglect
MeSH Terms: conditions — Stroke; Brain Injuries; Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Treatment (Experimental): Computerized Plasticity-based Adaptive Cognitive Training requiring a total maximum of 39 treatment sessions, 4-5 times weekly, ~30 mins each session.
  Interventions: Other: Computerized Plasticity-based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training requiring a total maximum of 39 treatment sessions, 4-5 times weekly, ~30 mins each session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-based Adaptive Cognitive Training — Computerized Plasticity-based Adaptive Cognitive Training requiring a total maximum of 39 treatment sessions, 4-5 times weekly, ~30 mins each session.
  Arms: Experimental Treatment
Other: Commercially available computerized training — Commercially available computerized training requiring a total maximum of 39 treatment sessions, 4-5 times weekly, ~30 mins each session.
  Arms: Active Comparator

SUMMARY:
Problems with attention are a common and debilitating consequence of brain injury. Studies show that poor attention is the number one predictor of poor cognitive functioning one year post-injury. This is due to the fact that attention is a necessary component of more complex cognitive functions such as learning & memory, multi-tasking and problem solving. In many cases, individuals may exhibit problems with spatial attention known as 'hemi-spatial neglect syndrome' or simply 'neglect'. Many studies now show that the processing machinery of the brain is plastic and remodeled throughout life by learning and experience, enabling the strengthening of cognitive skills or abilities. Research has shown that brief, daily computerized cognitive training that is sufficiently challenging, goal-directed and adaptive enables intact brain structures to restore balance in attention and compensate for disruptions in cognitive functioning. The study aims to understand how our computer program can affect cognition and attention in those with acquired brain injury.

DETAILED DESCRIPTION:
Following consent, participants will engage in an assessment process to determine eligibility. Once eligibility is confirmed, participants will be scheduled for another assessment session to determine current level of cognitive function. This process consists of paper-pencil surveys and computerized tests. Following the assessment process, participants will engage in an Internet browser-delivered training sessions conducted on any internet-accessible computer. The computerized training sessions can be done up to 7 times a week (once a day) or at participant's convenience (we recommend 5 times a week). Following the completion of training, the participant's cognitive function will be re-assessed and again after 3-month no-contact period. Participation is voluntary and participants may withdraw from the study at any time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of an acquired brain injury (which may be in the form of a stroke or brain tumor removal) and
* Evidence of deficit on at least 2 out of 4 assessment measures of Spatial Neglect: Mesulam Cancelation task (ages 50 and younger > 0 omissions; 51-80 > 4 omissions), Dual task (>19% difference in accuracy for right - left target trials), Tone Counting task (< 94% total accuracy), or Landmark task (deviation from objective center as determined by the 95% confidence interval, with neglect indicated with 'Y' and no neglect with 'N' following completion of task).
* Must be at least 3 months out from their most recent acquired brain injury, stroke, or brain tumor removal
* Fluent English speakers
* Adequate sensorimotor capacity to participate in the trial, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse

Exclusion Criteria:

* A conjunction of prior acquired brain injury and score >8 on Blessed Scale - Short Form
* Diagnosis of severe depression (a score of >29 on Beck Depression Inventory (BDI-II)
* Diagnosis of chronic psychiatric disorders with associated cognitive impairments, eg. Schizophrenia
* Diagnosis of illness, condition or treatment with known cognitive consequences, eg. chemotherapy
* Active Suicidal Ideation with Specific Plan and Intent or any suicide-related behaviors within 2 months of consent
* A current or significant past history of substance abuse
* Difficulty completing assessments and/or comprehending requirements of trial
* Enrollment in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device or behavioral treatment that could affect the outcome of this study
* Complete primary visual field deficit, score of 3 on NIH Stroke Scale - Visual Field Subscale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Performance on Posner Cueing Task | At 3 months
  Between-group magnitude of change in reaction time (RT) for RT detecting targets appearing on the left side of the display minus the RT for detecting targets appearing on the right side of the display as measured by Posner Cueing Task. Positive reaction time difference scores indicate a rightward bias; whereas, negative reaction time difference scores indicate a leftward bias in spatial attention.

SECONDARY OUTCOMES:
Change in Spatial Cognition (Multiple scores are aggregated to arrive at a single composite score) | At 3 months and at 6 months
  Between-group magnitude of change in composite score with the measure constructed from Greyscales Task (perceptual bias score) and Spatial Working Memory Task (percent accuracy for targets).
  The composite is composed of the individual measures combined as follows:
  i. For each included variable convert the distribution of raw scores in the Intent-to-Treat population at baseline to z-scores (with a mean of 0 and a standard deviation of 1).
  ii. Compute the average of all z-scores to create a single score for the composite measure.
Change in Cognitive Performance (Multiple scores are aggregated to arrive at a single composite score) | At 3 months and at 6 months
  Between-group magnitude of change in composite score with the measure constructed from Delis-Kaplan Executive Function System Verbal Fluency (Letter Fluency, raw scores; Category Fluency total, raw scores; Category Switching total, raw scores; Category Switching, switching Accuracy total, raw scores), Wechsler Adult Intelligence Scale (WAIS-IV) Digit Span total (sum of forward, backward, sequencing raw scores), WAIS-IV Digit Span (Forward total, raw scores; Backward total, raw scores; Sequencing total, raw scores), and Gradual Continuous Performance Task (percent accuracy for targets and standard deviation (SD) of average reaction time for non-targets).
  The composite is composed of the individual measures combined as follows:
  i. For each included variable convert the distribution of raw scores in the Intent-to-Treat population at baseline to z-scores (with a mean of 0 and a SD of 1).
  ii. Compute the average of all z-scores to create a single score for the composite measure.
Change in Functional Ability (Multiple scores are aggregated to arrive at a single composite score) | At 3 months and at 6 months
  Between-group magnitude of change in composite score with the measure constructed from Catherine Bergego Scale total (raw score) and Barthel Index total (raw score).
  The composite is composed of the individual measures combined as follows:
  i. For each included variable convert the distribution of raw scores in the Intent-to-Treat population at baseline to z-scores (with a mean of 0 and a standard deviation of 1).
  ii. Compute the average of all z-scores to create a single score for the composite measure.
Change in Quality of Life (Multiple scores are aggregated to arrive at a single composite score) | At 3 months and at 6 months
  Between-group magnitude of change in composite score with the measure constructed from SF-12v2 Health Survey Physical and Mental Component Scores.
  The composite is composed of the individual measures combined as follows:
  i. For each included variable convert the distribution of raw scores in the Intent-to-Treat population at baseline to z-scores (with a mean of 0 and a standard deviation of 1).
  ii. Compute the average of all z-scores to create a single score for the composite measure.
Change in Quality of Sleep: Pittsburgh Sleep Quality Index (Multiple scores are aggregated to arrive at a single composite score) | At 3 months and at 6 months
  Between-group magnitude of change in composite score with the measure constructed from Pittsburgh Sleep Quality Index (PSQI, sum of component scores), PSQI Sleep Efficiency (raw score), and PSQI Component scores.
  The composite is composed of the individual measures combined as follows:
  i. For each included variable convert the distribution of raw scores in the Intent-to-Treat population at baseline to z-scores (with a mean of 0 and a standard deviation of 1).
  ii. Compute the average of all z-scores to create a single score for the composite measure.
Performance on Posner Cueing Task | At 6 months
  Between-group magnitude of change in reaction time (RT) for RT detecting targets appearing on the left side of the display minus the RT for detecting targets appearing on the right side of the display as measured by Posner Cueing Task. Positive reaction time difference scores indicate a rightward bias; whereas, negative reaction time difference scores indicate a leftward bias in spatial attention.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Friedrich FJ, Egly R, Rafal RD, Beck D. Spatial attention deficits in humans: a comparison of superior parietal and temporal-parietal junction lesions. Neuropsychology. 1998 Apr;12(2):193-207. doi: 10.1037//0894-4105.12.2.193. PMID 9556766
- [Background] Husain M, Kennard C. Visual neglect associated with frontal lobe infarction. J Neurol. 1996 Sep;243(9):652-7. doi: 10.1007/BF00878662. PMID 8892067
- [Background] Heilman KM, Bowers D, Valenstein E, Watson RT. Disorders of visual attention. Baillieres Clin Neurol. 1993 Aug;2(2):389-413. No abstract available. PMID 8137006
- [Background] Mort DJ, Malhotra P, Mannan SK, Rorden C, Pambakian A, Kennard C, Husain M. The anatomy of visual neglect. Brain. 2003 Sep;126(Pt 9):1986-97. doi: 10.1093/brain/awg200. Epub 2003 Jun 23. PMID 12821519
- [Background] Posner MI, Walker JA, Friedrich FJ, Rafal RD. Effects of parietal injury on covert orienting of attention. J Neurosci. 1984 Jul;4(7):1863-74. doi: 10.1523/JNEUROSCI.04-07-01863.1984. PMID 6737043
- [Derived] Vleet TV, DeGutis J, Dabit S, Chiu C. Randomized control trial of computer-based rehabilitation of spatial neglect syndrome: the RESPONSE trial protocol. BMC Neurol. 2014 Feb 7;14:25. doi: 10.1186/1471-2377-14-25. PMID 24502769

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT01965951/SAP_001.pdf